CLINICAL TRIAL: NCT06220279
Title: Overall Comparison of Single Dose 100mg Rectal Diclofenac With Double Doses of 20mg Twelve Hours Apart Oral Diclofenac for Pain Relief Both for 24 Hours After Episiorrhahpy, Southeast Nigeria.
Brief Title: Efficacy of Single Dose Rectal Diclofenac With Oral Diclofenac for the Relief of Perineal Pain Within 24 Hours After Episiotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Teaching Hospital Abakaliki (Other Government)
Responsible Party: Principal Investigator, Nwali Matthew Igwe, Principal Investigator, Federal Teaching Hospital Abakaliki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRAEP2023CT
Record Dates: First submitted 2024-01-14; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Pain Relief After Episiotomy
MeSH Terms: interventions — Diclofenac

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1, oral diclofenac (Active Comparator): Two doses of 50mg oral diclofenac 12 hours apart was administered to this arm
  Interventions: Drug: Diclofenac
- Arm 2, rectal diclofenac (Active Comparator): 100mg diclofenac was administered rectally to this arm
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Diclofenac — Each were monitored for pain within 24 hours

SUMMARY:
Episiotomy is the commonest surgical procedure performed on parturient. It is usually associated with perineal pain which is particularly severe in the first 24 hours post repair. Perineal pain after episiorrhaphy if not adequately managed puts the woman into painful distress thus preventing good immediate post-partum care for the newborn. The aim is to compare the efficacy of single dose rectal diclofenac with oral diclofenac for the relief of perineal pain within 24 hours after episiotomy repair at Alex Ekwueme Federal University Teaching Hospital Abakaliki.

DETAILED DESCRIPTION:
Episiotomy is the commonest surgical procedure performed on parturient. It is usually associated with perineal pain which is particularly severe in the first 24 hours post repair. Perineal pain after episiorrhaphy if not adequately managed puts the woman into painful distress thus preventing good immediate post-partum care for the newborn.

Aim: To compare the efficacy of single dose rectal diclofenac with oral diclofenac for the relief of perineal pain within 24 hours after episiotomy repair at Alex Ekwueme Federal University Teaching Hospital Abakaliki.

Materials and Methods: This was a randomized controlled trial that involved 146 women that had episiorrhaphy between June and December 2020. The women were randomized into two groups of 73 women each using computer generated random numbers. One group received 100mg of diclofenac suppository stat while the other group received 2 doses of 50mg of oral diclofenac 12 hours apart, both for 24 hours after episiorrhaphy. Pain was assessed at 1, 4, 8, 16 and 24 hours post episiorraphy using a Visual Analogue Scale. Maternal satisfaction for the mode of the pain relief was assessed using the Likert scale after 24 hours. Data obtained was analyzed using Statistical Package for Social Science software version 25.

The perineal pain was categorized into: no pain (0cm), mild (1-3cm), moderate (4-7cm) and severe (8-10cm), while maternal satisfaction was categorized into: Very satisfied, Satisfied, Neutral, Dissatisfied, Very dissatisfied. Categorical variables were summarized using frequencies and proportion. Quantitative variables were summarized with means and standard deviation. Student t-test was used for comparison between the group means for continuous variables while Chi-squared test was used to compare categorical variables. Statistical significance was obtained when p-value was ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Uncomplicated pregnancy
* Gestational age of 37 weeks and above who had episiotomy
* Singleton gestation
* Vaginal delivery
* Instrumental vaginal delivery
* Consented women

Exclusion Criteria:

* Women that declined consent
* Postpartum hemorrhage.
* Women who had perineal tear
* History of peptic ulcer diseases
* History of bleeding coagulopathies
* Adverse reaction or hypersensitivity to diclofenac
* Any woman with special postpartum pain relief plan such as sickle cell disease patient
* Preeclamptic/eclamptic, renal and liver diseases patients.
* Parturient on epidural anesthesia

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Adequate pain relief after drug administration | 24hours
  Clients satisfaction

CONTACTS AND LOCATIONS:
Locations (2):
- Nigeria (2):
  - Alex Ekwueme Federal University Teaching Hospital, Abakaliki, Ebonyi State
  - Federal Teaching Hospital, Abakaliki, Abakaliki, Ebonyi State

IPD SHARING:
Plan to Share IPD: No